CLINICAL TRIAL: NCT01742676
Title: A Single Center, Open-label, Randomized Pilot Study to Evaluate the Safety and Efficacy of Modified-release Tacrolimus, ADVAGRAF®, Versus Those of Twice-daily Tacrolimus, PROGRAF®, in Stable Renal Recipients (SINGLE)
Brief Title: A Single Center, Open-label, Randomized, Pilot Study to Evaluate the Safety and Efficacy of a Tacrolimus Modified Release, ADVAGRAF®, Versus Tacrolimus Twice Daily, PROGRAF® in Stable Renal Recipients
Acronym: SINGLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADV-KT-03
Record Dates: First submitted 2012-12-04; First posted 2012-12-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Renal Transplantation; Kidney Transplantation; Stable Renal Recipients
Keywords: tacrolimus; kidney
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADVAGRAF group (Experimental)
  Interventions: Drug: ADVAGRAF
- PROGRAF group (Active Comparator)
  Interventions: Drug: PROGRAF

INTERVENTIONS:
Drug: ADVAGRAF — oral
  Other Names: modified release tacrolimus
  Arms: ADVAGRAF group
Drug: PROGRAF — oral
  Other Names: twice-daily tacrolimus
  Arms: PROGRAF group

SUMMARY:
The purpose of this study is to evaluate and compare the safety and efficacy of two drugs (ADVAGRAF® and PROGRAF® groups) in patients who received renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

Only patients who meet the following inclusion criteria should be enrolled.

1. Patients who received a kidney at least within 12 months of their study enrollment (from a deceased or living donor)
2. Patients whose tacrolimus dose have not been changed in at least 12 weeks from their study enrollment and whose minimum blood tacrolimus concentration mean value is within 3-10 ng/ml
3. Female patients who showed a negative result in the serum pregnancy test and who agreed to use an effective contraceptive method during the study period
4. Patients who are clinically stable based on the judgment of the investigator
5. Patients who were given enough information regarding the study, understood the objectives and risks of the study, and signed the informed consent form

Exclusion Criteria:

Patients who fall under any of the following criteria should not be enrolled in this study.

1. Patients who had received any other organ except a kidney
2. Patients who showed an acute rejection reaction within 12 weeks of their enrollment or who showed an acute rejection reaction that required antilymphocyte antibody therapy within 24 weeks
3. Patients who were diagnosed with a newly developed malignant tumor (Patients with successfully treated squamous cell/basal cell carcinoma can be enrolled, though.)
4. Patients who have a known allergy to the investigational drug (the test/control drug) or to tacrolimus
5. Patients who have an unstable medical condition that may affect the evaluation of the study's objectives based on the investigator's judgment
6. Patients who have any form of drug abuse or mental illness that might complicate communication with the investigators based on the investigator's judgment
7. Patients who are currently participating in another clinical trial or who received the investigational drug in another trial within 28 days of their enrollment
8. Patients who are receiving prohibited concomitant medications or who received those medications within 28 days of their enrollment
9. Patients who are pregnant or breastfeeding
10. Patients who had been HIV-positive
11. Patients who are considered non-compliant with the scheduled study visits in the protocol
12. Patients who have abnormal kidney functions or a serum creatinine level higher than 1.6 mg/dL/GFR (MDRD) or less than 30 mL/min at the screening visit
13. Patients who have "Creeping creatinine" (a 20% increase in their creatinine for six months before their enrollment)
14. Patients who have abnormal liver functions: i.e., whose SGPT/ALT and/or SGOT/AST and/or bilirubin is twice higher than the normal range in the center, and who have liver cirrhosis
15. Patients who have an underlying disease such as focal segmental glomerulosclerosis (FSGS) or type II membranoproliferative glomerulonephritis (Type II MPGN)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | at 24 weeks

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | at 24 weeks
  Calculated by Modification of Diet in Renal Disease equation
Incidence of rejection reactions | at 24 weeks
Blood pressure | at 24 weeks
Survival rate of the grafts | at 24 weeks
Subject's physical condition (SF-35) | at 24 weeks
  Evaluation of subject's physical condition

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Seoul, South Korea